CLINICAL TRIAL: NCT01036659
Title: Evaluation of Ecallantide for Acute Treatment of Angiotensin Converting Enzyme Inhibitor Induced Angioedema
Brief Title: Evaluation of Ecallantide for the Acute Treatment of Angiotensin Converting Enzyme Inhibitor Induced Angioedema
Acronym: ACE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bernstein, Jonathan A., M.D. (Individual)
Collaborators: Dyax Corp. (Industry)
Responsible Party: Jonathan a. Bernstein, M.D., UC Physicians, Department of Internal Medicine Division of Immunology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACE Induced Angioedema
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Angioedema
Keywords: acute angiotensin converting enzyme inhibitor angioedema
MeSH Terms: conditions — Angioedema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ecallantide in conjunction with Conventional Therapy (Active Comparator)
  Interventions: Drug: ecallantide - Kallikrein inhibitor that blocks the production of bradykinin
- Conventional therapy and placebo (Placebo Comparator)
  Interventions: Drug: ecallantide - Kallikrein inhibitor that blocks the production of bradykinin
- Historical Evaluation (No Intervention)

INTERVENTIONS:
Drug: ecallantide - Kallikrein inhibitor that blocks the production of bradykinin — subcutaneous dose of 30mg of ecallantide or placebo (three 10 mg SC injections at three different sites ((arms, legs, abdomen). Injections are not to be administered at the attack location.
  Arms: Conventional therapy and placebo; Ecallantide in conjunction with Conventional Therapy

SUMMARY:
The investigators will conduct a double-blind, randomized controlled trial comparing the safety and effectiveness of ecallantide to conventional therapy. A rescue cross-over design will be used such that patients failing to improve on standard therapy will additionally be treated with ecallantide. Therefore, a historical control cohort will be enrolled for analysis of secondary endpoints. In addition, since some patients treated with conventional therapy may improve rapidly and therefore not be eligible for inclusion in the study, the investigators will enroll these patients as an observational arm to enable the conduct of sensitivity analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of any race or ethnicity 18 or older. The locations of the study will permit all racial and ethnic distribution in the study
2. Must currently be on an ACE inhibitor
3. Presenting with ACE induced angioedema within 12 hours after onset. This is to be documented in the source document and CRF
4. All females of childbearing age must have a negative pregnancy test prior to administration of the study drug.

Exclusion Criteria:

1. Participation in another investigational study within 30 days prior to enrollment
2. Patients who improve on conventional (standard of care) therapy
3. Patients previously treated with ecallantide
4. Hypersensitivity to ecallantide
5. Pregnancy or breast feeding
6. Other definable causes of angioedema (i.e., hereditary or acquired angioedema)
7. Patients receiving C-1 inhibitor as prophylaxis
8. Treatment requiring tranexamic acid, and epsilon-aminocaproic acid
9. Receiving fresh frozen plasma within 3 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Objective criteria that allow for discharge directly from the ED at or before 4 hours:(stable vital signs, no evidence of stridor, dysphagia or drooling, edema has regressed to or did not progress beyond Class I. | 18 months

SECONDARY OUTCOMES:
Time to meet objective discharge criteria, Physician assessment of angioedema improvement measured using the Symptom Complex Response Assessment at 2 hours post-treatment and 4 hours post-treatment. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A. Bernstein, M.D., Principal Investigator — UC Physicians, Division of Immunology; Joseph Moellman, MD, Principal Investigator — UC Physicians, Department of Emergency Medicine
Locations (3):
- United States (3):
  - The Jewish Hospital, Cincinnati, Ohio
  - Univeristy Hospital, Cincinnati, Ohio
  - UC Physicians, Dpt of Internal Medicine, Division of Immunology, Cincinnati, Ohio

REFERENCES:
- [Derived] Bernstein JA, Moellman JJ, Collins SP, Hart KW, Lindsell CJ. Effectiveness of ecallantide in treating angiotensin-converting enzyme inhibitor-induced angioedema in the emergency department. Ann Allergy Asthma Immunol. 2015 Mar;114(3):245-9. doi: 10.1016/j.anai.2014.12.007. Epub 2015 Jan 16. PMID 25601538